CLINICAL TRIAL: NCT05193071
Title: Early Antiplatelet for Minor Stroke Following Thrombolysis (EAST): a Prospective, Random, Double Blinded and Multi-center Study
Brief Title: Early Antiplatelet for Minor Stroke Following Thrombolysis (EAST)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Head of Neurology, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: y (2021) 109
Record Dates: First submitted 2021-12-31; First posted 2022-01-14 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Ischemic Stroke
Keywords: thrombolysis; minor stroke; early antiplatelet
MeSH Terms: conditions — Ischemic Stroke | interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- double antiplatelet group (Experimental): aspirin 100mg plus clopidogrel 300mg
  Interventions: Drug: Aspirin 100mg; Clopidogrel 300mg
- control group (Placebo Comparator): aspirin placebo plus clopidogrel placebo
  Interventions: Drug: Aspirin 100mg; Clopidogrel 300mg

INTERVENTIONS:
Drug: Aspirin 100mg; Clopidogrel 300mg — Aspirin 100mg plus Clopidogrel 300mg will be orally administrated after randomization

SUMMARY:
The current guideline recommends to give antithrombotic treatment 24 hours after intravenous thrombolysis in acute ischemic stroke. However, early neurological deterioration will occur in some patients due to no antithrombotic treatment, which is closely associated with poor outcome. The current trial aims to investigate the effectiveness and safety of early antithrombotic treatment after intravenous thrombolysis in minor stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old;
* Acute ischemic stroke patients who received intravenous thrombolysis within 4.5 hours of onset;
* NIHSS ≤ 5 within 6 hours after the end of intravenous thrombolysis, and no bleeding transformation was found in head CT examination;
* Premorbid mRS ≤ 1;
* Signed informed consent.

Exclusion Criteria:

* Premorbid mRS≥2;
* Uncontrolled severe hypertension (systolic pressure >180 mmHg or diastolic pressure >110 mmHg after drug treatment);
* Antithrombotic treatment within 24 hours before randomization;
* Significant dysphagia and inability to take the experimental drug orally;
* Allergy or contraindication to study drugs;
* Comorbidity with any serious diseases and life expectancy is less than half a year;
* Participating in other clinical trials within three months;
* Patients not suitable for this clinical study considered by researcher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1022 (Actual)
Dates: Start 2022-07-08 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-10-25 (Actual)

PRIMARY OUTCOMES:
The proportion of excellent prognosis | Day 90
  excellent prognosis is defined as modified Rankin Score (mRS) 0-1. The minimum and maximum values of mRS are 0 and 6, respectively; higher score mean a worse outcome

SECONDARY OUTCOMES:
The proportion of favorable prognosis | Day 90
  Favorable prognosis is defined as modified Rankin Score (mRS) 0-2. The minimum and maximum values of mRS are 0 and 6, respectively; higher score mean a worse outcome.
Distribution of modified Rankin Score (mRS) | Day 90
  The minimum and maximum values of mRS are 0 and 6, respectively; higher score mean a worse outcome.
Changes in National Institute of Health stroke scale (NIHSS) | 24 hours, 48 hours, and 10 days
  the minimum and maximum values of NIHSS are 0 and 42, respectively; higher NIHSS mean a worse outcome.
Occurrence of early neurologyical deterioration (END) | 24 hours
  END is defined as more than 2 point increase, but not result of cerebral hemorrhage, compared with baseline at 24 hours
The incidence of symptomatic intracerebral hemorrhage | 36 hours
  any evidence of bleeding on the head CT scan associated with clinically significant neurological deterioration (NIHSS score ≥4 points increase)
The incidence of any intracerebral hemorrhage | 36 hours
  the evidence of bleeding on the head CT or MRI scan
The incidence of stroke recurrence and other vascular events | Day 90
The death due to any cause | Day 90

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Hui-sheng Chen, Shenyang, None Selected
  - Department of Neurology, General Hospital of Northern Theater Command, Shenyang

IPD SHARING:
Plan to Share IPD: Undecided